CLINICAL TRIAL: NCT00695851
Title: A Phase I Randomized Dose-Seeking Trial of PCK3145 in Asymptomatic, Castrate Metastatic Prostate Cancer Patients.
Brief Title: Dose-Seeking Trial of PCK3145 in Asymptomatic, Castrate Metastatic Prostate Cancer Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ambrilia Biopharma, Inc. (Industry)
Responsible Party: Susan Slovin, MD, Memorial Sloan-Kettering Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-019
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Prostate Cancer
Keywords: PCK3145; Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tigapotide

ARMS (2):
- 1 (Experimental): 15 mg/m2 weekly of PCK3145
  Interventions: Drug: PCK3145
- 2 (Experimental): 7.5 mg/m2 twice per week of PCK3145
  Interventions: Drug: PCK3145

INTERVENTIONS:
Drug: PCK3145 — i.v. bolus either 15 mg/m2 weekly of PCK3145.
  Arms: 1
Drug: PCK3145 — by i.v. bolus 7.5 mg/m2 twice per week of PCK3145
  Arms: 2

SUMMARY:
The purpose of this study is to find out whether giving a drug called PCK3145 can reduce the level of a protein in the blood called MMP-9 as well as to find out how long the drug will remain in your system over time. This drug has been tested previously in prostate cancer patients abroad and has been shown to be safe with minimal side effects. However, we do not know whether changes in MMP-9 levels correlate with tumor shrinkage or symptom improvement. We would also like to evaluate the potential pain relief (analgesic) effect of PCK3145 at 15mg/m² i.v. weekly for 12 weeks on patients with both symptomatic and asymptomatic castrate metastatic prostate cancer who are dependent on opioid analgesics. We would also like to monitor pain through a brief pain questionaire, and determine the impact on markers of bone turnover.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have castrate metastatic prostate cancers are eligible based on the following criteria.
* Patients with prostate cancer must have castrate metastatic disease (i.e. disease progression following castration or treatment with a gonadotropin releasing hormone analog. Patients with prostate cancer may have progressing metastatic disease on imaging studies (bone scan, CT scan or MRI) in addition to a rising PSA.
* Biochemical progression will be defined as: A minimum of three rising PSA values from a baseline that are obtained 1 week or more apart, or two rising PSA values more than one month apart, where the percentage increase over the range of values is at least 25%.
* Maintaining castrate status: Patients who have not undergone surgical orchiectomy should continue on medical therapies [i.e. gonadotropin releasing hormone analogs] to maintain castrate levels of serum testosterone. Patients who are receiving an anti-androgen as part of first line hormonal therapy must have shown progression of disease off the anti-androgen prior to enrollment.
* Histologically confirmed diagnosis of prostate cancer per MSKCC review.
* No limitations on the duration of or number of prior therapies.
* Age ≥ 18 years
* Karnofsky performance status ≥ 70% (ECOG ≤ 1.0).
* Life expectancy of greater than 6 months.
* Hematologic: WBC ≥ 3000K/μl.
* Absolute neutrophil count ≥ 1500 K/μl
* Platelet count ≥ 100,000 K/μl.
* Hepatic: Total Bilirubin - within normal institutional limits
* AST < 1.5 x ULN, ALT < 1.5 x ULN.
* Renal: Creatinine < 2.0 or creatinine clearance > 55 mL/min
* Coagulation: Prothrombin time - Less than or equal to the ULN (upper limit of normal) unless patient is taking anticoagulants
* Patients must have recovered from the acute toxicities of any prior therapy, and not received chemotherapy, radiation therapy or other investigational anticancer therapeutic drugs for at least 4 weeks prior to entry.
* Ability to understand and the willingness to sign a written informed consent document.
* Testosterone < 50 ng/dl
* Patients may be symptomatic and must be dependent on opioid analgesics or nonsteroidal anti-inflammatory drugs

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from the adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with active brain metastases or epidural disease
* Uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* No current therapy with alternative/complementary drugs such as PC Plus, saw palmetto or Zyflamend.
* No rectal bleeding except that seen following radiation proctitis or known history of hemorrhoids.
* Non-prostate primary carcinoma except for non-melanoma skin cancer within previous 5 years.
* No uncontrolled cardiac arrhythmias.
* Patient taking steroids for cord compression or pain control are excluded. Patient on steroids for chronic conditions such as arthritis or asthma or on chronic hydrocortisone post ketoconazole will be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To explore the PK profiles and their association with two dosing schedules of PCK3145 given iv bolus in patients with asymptomatic castrate metastatic prostate cancer. | conclusion of the study

SECONDARY OUTCOMES:
To explore the association of 2 dosing schedules of PCK3145 with MMP-9 levels in asymptomatic pts with castrate metastatic prostate cancer. The results of this analysis will be used to establish a dose on which to build a phase II randomized trial. | conclusion of the study
To assess the safety and toxicity of PCK3145 at a dose of 150mg/m² i.v. bolus given weekly for 16 weeks. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org